CLINICAL TRIAL: NCT01749241
Title: Loteprednol Etabonate Ophthalmic Ointment vs. Soothe Night Time Ointment for Inflammation Following Eyelid Surgery
Brief Title: Efficacy of Loteprednol Ointment Following Eyelid Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participant enrolled
Sponsor: University of California, San Diego (Other)
Collaborators: Shiley Eye Center (Other); Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Bobby Korn, MD, PhD, Associate Professor of Ophthalmology, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BL31929
Record Dates: First submitted 2012-12-10; First posted 2012-12-13 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Post-operative Healing Following Blepharoplasty and Ptosis Repair

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loteprednol etabonate ointment (Experimental): This is the arm which contains loteprednol steroid
  Interventions: Drug: Loteprednol etabonate ophthalmic ointment
- Vehicle Ointment (Other): This arm contains vehicle only.
  Interventions: Drug: Vehicle Ophthalmic Ointment

INTERVENTIONS:
Drug: Loteprednol etabonate ophthalmic ointment — Thin ribbon ointment to assigned eye twice daily for 14 days
  Other Names: Lotemax ophthalmic ointment
  Arms: Loteprednol etabonate ointment
Drug: Vehicle Ophthalmic Ointment — Thin ribbon ointment to assigned eye twice daily for 14 days
  Arms: Vehicle Ointment

SUMMARY:
Inflammation occurs after any type of incisional surgery. This study will evaluate the efficacy of Loteprednol etabonate ointment vs. Soothe ointment (vehicle) for postoperative inflammation after routine eyelid surgery.

DETAILED DESCRIPTION:
Eyelid surgery such as blepharoplasty is often performed for functional and cosmetic indications. Following any incisional surgery, postoperative inflammation occurs at the surgical site. This study will evaluate the efficacy of reducing postoperative inflammation after bilateral eyelid surgery using Loteprednol etabonate (steroid) vs. Soothe ointment (vehicle of Loteprednol etabonate). Common postoperative changes at the incision include: erythema, thickening/elevation of the skin, pigmentary changes and pain. The use of a topically applied steroid would be expected to reduce inflammation and this study will evaluate this. For each patient, one eyelid will be randomly chosen to treat with medication and the other eyelid will be treated with vehicle ointment and by using the same patient, each patient will be internally controlled. Antibiotic prophylaxis is often given after eyelid surgery and this will be used in all patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Scheduled for bilateral eyelid surgery
* Willing and able to return for all study visits
* Willing and able to administer treatments as required
* Understand and sign informed consent approved by UCSD institutional review board

Exclusion Criteria:

* History of allergy to investigational drug (Loteprednol etabonate) or ingredient in drug including petrolatum
* History of collagen vascular disease and receiving concurrent treatment that could interfere with interpretation of study results
* Concurrent ocular therapy with nonsteroidal anti-inflammatory drugs, mast cell stabilizers, antihistamines, decongestants, immunosuppresants, and systemic or ocular corticosteroids
* History of immunodeficiency
* Prior eyelid or facial surgery
* Prior ocular or orbital trauma
* History of ocular hypertension, steroid responder, or glaucoma
* Pregnancy or lactation
* Uncontrolled systemic disease or significant illness
* Any other condition the investigator believe would pose a significant hazard to the subject if the investigational therapy were initiated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Inflammation | 24 weeks after surgery
  Inflammatory changes of the periocular skin will be assessed by several criteria including: 1. Erythema 2. Wound elevation 3. Pigmentary changes 4. Exudate 5. Excoriation 6. Crusting 7. Scaling 8. Pain 9. Itching

CONTACTS AND LOCATIONS:
Overall Officials: Bobby Korn, MD PhD, Principal Investigator — UCSD Med
Locations (1):
- Shiley Eye Center, La Jolla, California, United States

REFERENCES:
- [Result] Comstock TL, Paterno MR, Singh A, Erb T, Davis E. Safety and efficacy of loteprednol etabonate ophthalmic ointment 0.5% for the treatment of inflammation and pain following cataract surgery. Clin Ophthalmol. 2011;5:177-86. doi: 10.2147/OPTH.S16832. Epub 2011 Feb 10. PMID 21383946
- [Result] A double-masked, placebo-controlled evaluation of 0.5% loteprednol etabonate in the treatment of postoperative inflammation. The Loteprednol Etabonate Postoperative Inflammation Study Group 2. Ophthalmology. 1998 Sep;105(9):1780-6. doi: 10.1016/s0161-6420(98)99054-6. PMID 9754192